CLINICAL TRIAL: NCT05871216
Title: Evaluation of Functional Instability Using the "Delos Proprioceptive System" in Patients Suffering From Collagen Disease and Joint Hypermobility
Brief Title: Functional Instability in Patients Suffering From Collagen Disease and Joint Hypermobility
Acronym: VIPIA
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 0006530
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hypermobility Syndrome; Danlos Disease, Ehlers; Collagen Diseases; Joint Hypermobility; Laxity of Ligament
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Collagen Diseases; Joint Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Joint Hypermobility Syndrome: Patients suffering from Joint Hypermobility Syndrome with a moderate/severe degree of joint hypermobility (Beighton-Horan Joint Mobility Index score 3-9)
  Interventions: Diagnostic Test: Clinical tests and balance evaluation using the Delos Proprioceptive System

INTERVENTIONS:
Diagnostic Test: Clinical tests and balance evaluation using the Delos Proprioceptive System — Each patient is evaluated using clinical tests (Time up and go test, 6 minutes walking test), scales (BORG scale, Beighton score), and the ''Delos Proprioceptive System'' to assess balance control and proprioception with bipodalic and monopodalic tests.

SUMMARY:
A joint is considered "hypermobile" when it has a greater range of motion than normal for a given age, ethnicity or gender. Many people have asymptomatic hyperlaxity in multiple joints, a condition called Generalized Joint Hypermobility (GJH).

Conversely, hyperlaxity can be symptomatic, a condition that has been defined "Joint Hypermobility Syndrome" - JHS.

Diagnosis of JHS is commonly performed by applying the revised Brighton criteria. Based on these criteria, an individual is diagnosed with JHS with a Beighton score >/= 4/9, and arthralgia for 3 or more months in 4 or more joints (major criteria).

The dynamic body balance test (i.e. the stability test with multiple single-leg jumps) can provide information regarding the effectiveness of the feedforward and feedback mechanisms in correcting the postural deviations necessary to achieve successful performance during daily and sporting activities. Such assessment may also be useful to demonstrate deficiencies in balance, especially in young patients with increased physical activity.

The aim of this study is to examine the postural balance of individuals with JHS by performing stability tests in monopodalic and bipodalic stance with the "Delos Postural Proprioceptive System"

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate (Beighton-Horan Joint Mobility Index score from 3 to 4) or severe (Beighton-Horan Joint Mobility Index score from 5 to 9) joints hyperlaxity at the clinical evaluation

Exclusion Criteria:

* Obesity (BMI > 25) and weight > 90 kg
* Practice of competitive sport
* Orthopedic (complex surgery of the spine and lower limbs), neurological (spasticity, stroke), and oncological comorbidities
* Orthostatic / walking inability
* Absence of joints hyperlaxity at the clinical evaluation (Beighton-Horan Joint Mobility Index score from 0 to 2)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with moderate (Beighton-Horan Joint Mobility Index score from 3 to 4) or severe (Beighton-Horan Joint Mobility Index score from 5 to 9) joints hyperlaxity at the clinical evaluation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessing proprioception and postural control | baseline
  Assessing proprioception and postural control using the Delos Proprioceptive System to obtain static and dynamic stability indicators

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS-Istituto Ortopedico Rizzoli, Bologna, Italy